CLINICAL TRIAL: NCT04405219
Title: Preoperative Smoking Cessation, Preoperative Anxiety, Postoperative Anxiety and Pain Relationship
Brief Title: Smoking Cessation, Anxiety, Pain Relationship
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Arzu Esen Tekeli, Assistant Professor Doctor, Yuzuncu Yil University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2018/05
Record Dates: First submitted 2020-05-18; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Smoking Cessation; Anxiety; Pain
Keywords: Smoking Cessation; anxiety; pain; VAS Scores; STAI Values
MeSH Terms: conditions — Smoking Cessation; Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- smokers (S) (Sham Comparator)
  Interventions: Other: The Relationship Between Preoperative Smoking Cessation, Anxiety, Pain
- non smokers (NS) (Active Comparator)
  Interventions: Other: The Relationship Between Preoperative Smoking Cessation, Anxiety, Pain

INTERVENTIONS:
Other: The Relationship Between Preoperative Smoking Cessation, Anxiety, Pain — Preoperative anxiety high score suggests stress related to surgery and anesthesia. High anxiety scores independent of post-operative pain showed smoking withdrawal.

SUMMARY:
Smoking, anxiety and pain are clearly related conditions. We aimed to reveal the relationship between smoking cessation before surgery and preoperative anxiety, postoperative anxiety and pain in chronic smokers.

METHODS ASA I-II group patients without chronic disease and history of drug use were included in the study. Those who did not want to participate in the study, patients with ASA III and above were excluded from the study. The patients were randomized into 2 groups: smokers (Group S, n = 60) and non-smokers (Group NS, n = 60). Group S was asked to quit smoking 2 weeks before the operation. Preoperative period and postoperative 0, 2, 4. And 6. hour Spielberger State-Trait Anxiety Inventory (STAI) values, postop 0., 2., 4., 6. hour Visual Analogue Scale (VAS) values were recorded.

DETAILED DESCRIPTION:
it has been revealed in the current study that smoking, pain and anxiety are interrelated with each other. In the preoperative period, high anxiety scores are related to surgery and anesthesia stress. High anxiety scores in the smoker group both in the preoperative period and in the postoperative period are associated with smoking cessation. While the pain scores were similar in the postoperative period, high anxiety scores strengthened the idea of smoking withdrawal and this study gained value. We believe that future studies with a large number of patients, with different parameters and multiple centers will strengthen the results.

ELIGIBILITY:
Inclusion Criteria:

* ASA I,II patients
* planned Rhinoplasti cases
* accepted participating study

Exclusion Criteria:

* Patients with chronic systemic disorders,
* ASA III and above situation
* emergency and bleeding cases,
* patients with any cardiac and neurological disorders,
* refused to participate in the study

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2018-02-17 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
Anxiety | 2 hours
  assesed with STAI form

SECONDARY OUTCOMES:
pain scores | 2 hours
  independent of anxiety, assesed with VAS scores

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Esen Tekeli, MD, Principal Investigator — yuzuncu yil
Locations (2):
- Turkey (Türkiye) (2):
  - Van Yuzuncu Yil University Faculty of Medicine Department of anesthesiology and reanimation, Van, Tuşba
  - Van Yuzuncu Yil University, Van, Tuşba

IPD SHARING:
Plan to Share IPD: Undecided
I do not want to share before publishing